CLINICAL TRIAL: NCT00926081
Title: Exercise Training Versus Best Medical Treatment Only in Peripheral Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Oliver Schlager, Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK056/2007
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2011-12

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Artery Disease; Quality of Life; Outcome; Endothelial Progenitor Cells; Microcirculation
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Best medical treatment (No Intervention): Patients with peripheral artery disease receiving best medical treatment only
- Supervised exercise training (Active Comparator): Patients with peripheral artery disease receiving best medical treatment plus supervised exercise training
  Interventions: Behavioral: Supervised exercise training

INTERVENTIONS:
Behavioral: Supervised exercise training — A standardized supervised exercise training program
  Other Names: Standardized supervised exercise training
  Arms: Supervised exercise training

SUMMARY:
The aim of the investigators' study is to analyze the value of supervised exercise training combined with medical therapy versus best medical treatment only with respect to quality of life. Furthermore, the investigators aim to evaluate the effect of supervised exercise training on microcirculation, peripheral endothelial progenitor cells as well as on future major cardiovascular adverse events.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) affects 7 - 12% of the population aged over 50 years. Over an age of 60 years up to 20% are suffering from PAD in Western societies. Both, percutaneous transluminal angioplasty (PTA) and surgical repair (bypass graft, thrombectomy) are well established procedures to improve peripheral arterial perfusion. However, long-term results remain disappointing: Low patency-rates are associated with clinical deterioration. Moreover, clinical outcome is often limited by early major cardiovascular adverse events (myocardial infarction, stroke).

Therefore, medical therapy plays a major role in the management of PAD patients: Antihypertensive medication, statins as well as an adequate diabetes therapy are important cornerstones in the therapeutical management of PAD. Prior studies have shown that regular supervised exercise training can improve patients´walking impairment.

We hypothesize that regular supervised exercise training significantly improves Quality of Life and decreases the occurence of future major cardiovascular adverse events. We further aim to investigate the effect of exercise training on peripheral microcirculation and endothelial progenitor cells.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral artery disease with intermittent claudication (Rutherford 2-3)
* Exercise tolerance
* Ankle brachial index < 0,9
* Ability to life independently at home

Exclusion Criteria:

* No PAD
* Asymptomatic PAD
* Ischemic rest pain
* Exercise tolerance limited by other factors than claudication (e.g., coronary artery disease, dyspnoea, poorly controlled blood pressure, any kind of restriction of the musculoskeletal system which might have an influence on the efficiency of exercise training)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | 1 year

SECONDARY OUTCOMES:
Endothelial progenitor cells | 1 year
Inflammatory parameters | 1 year
Ankle brachial index | 1 year
Pain-free walking distance | 1 year
Peripheral transcutaneous oxygen pressure | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Steiner-Boeker, MD, Principal Investigator — Department of Angiology, Medical University Vienna
Locations (1):
- Department of Angiology, Vienna Medical University, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Schlager O, Hammer A, Giurgea A, Schuhfried O, Fialka-Moser V, Gschwandtner M, Koppensteiner R, Steiner S. Impact of exercise training on inflammation and platelet activation in patients with intermittent claudication. Swiss Med Wkly. 2012 Aug 14;142:w13623. doi: 10.4414/smw.2012.13623. eCollection 2012. PMID 22893497